CLINICAL TRIAL: NCT07379203
Title: A Phase 2b Randomised Placebo Controlled Trial of Valganciclovir for Cytomegalovirus Viraemia in Adults and Adolescents With Advanced HIV Disease
Brief Title: ValgaNciclovIR for CMV Viraemia in AdvaNced HIV diseAse
Acronym: NIRVANA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other); London School of Hygiene and Tropical Medicine (Other); St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIRVANA
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cytomegalovirus (CMV) Infection
Keywords: Cytomegalovirus; Advanced HIV disease; valganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valganciclovir (Experimental): Valganciclovir 900mg daily for 28 days
  Interventions: Drug: Valganciclovir
- Arm B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir
  Arms: Valganciclovir
Drug: Placebo — Placebo
  Arms: Arm B

SUMMARY:
The goal of this clinical trial is to learn if valganciclovir works to treat cytomegalovirus (CMV) infection in people with advanced HIV disease. It will also look at the safety of valganciclovir and how the body handles the drug.

The main questions this study aims to answer are:

Does valganciclovir safely lower the amount of CMV virus in the blood of people with advanced HIV disease?

What medical problems or side effects do participants have when taking valganciclovir?

Researchers will compare valganciclovir to a placebo (a look-alike tablet that does not contain any active drug) to see if valganciclovir works better than no treatment for CMV.

Who can take part

Adults and adolescents (15 years and older) who:

Are living with HIV

Have a CD4 count of 100 or less (meaning their immune system is very weak)

Have CMV detected in their blood

People who are pregnant, breastfeeding, very unwell, or have certain blood or kidney problems cannot take part.

What will happen in the study

Participants will:

Be randomly assigned (like flipping a coin) to take either valganciclovir 900 mg or a placebo once a day for 4 weeks

Continue to receive standard medical care for HIV and any other infections

Be followed for 12 weeks after starting the study treatment

During this time, participants will:

Have blood tests to check CMV, HIV, and general health

Have regular medical check-ups (daily in hospital, then at weeks 1, 2, 3, 4, 8, and 12)

Be monitored closely for side effects, such as low blood counts or kidney problems

Why this study is important

Even though HIV treatment is widely available, many people still come to hospital with advanced HIV disease. In this group, about one in five people die despite starting antiretroviral therapy (ART). Reactivation of CMV is very common in these patients and has been linked to a higher risk of death.

Valganciclovir is a medicine that stops CMV from multiplying. If it proves to be safe and effective in this study, it could become part of routine care to help reduce deaths in people with advanced HIV disease.

Study design

Type: Phase 2b, double-blind, randomised, placebo-controlled trial

Sites: Helen Joseph Hospital (South Africa) and Mulago National Referral Hospital (Uganda)

Number of participants: 150 (130 in the main trial, 20 in a smaller sub-study)

Duration: Each participant will be followed for 12 weeks; total study duration about 2 years

Possible risks and benefits

Risks: Valganciclovir can cause low white blood cells, anaemia, or low platelets. These effects will be checked for regularly, and treatment will be stopped if unsafe levels are found.

Benefits: The study may or may not directly benefit participants. However, it could provide important information that helps improve care for people with advanced HIV disease in the future.

Oversight and safety

The study is being conducted by researchers in Uganda, South Africa, the UK, and the USA, and follows international Good Clinical Practice (GCP) guidelines.

An independent Data Safety and Monitoring Committee (DSMC) will regularly review safety information to protect participants.

DETAILED DESCRIPTION:
Scientific Background and Rationale

Despite the widespread availability of antiretroviral therapy (ART), approximately 30 percent of adults with HIV continue to present to care with AHD, defined as a CD4 count < 200 cells/μL or a World Health Organization (WHO) stage 3 or 4 disease. In sub-Saharan Africa, mortality among hospitalised adults with AHD remains unacceptably high, typically exceeding 20 percent within weeks of admission. There is an urgent need for interventions that reduce early mortality in this extremely vulnerable population.

Cytomegalovirus is a ubiquitous herpesvirus that remains latent after primary infection but can reactivate when immunity is impaired. In individuals with AHD, CMV reactivation is common: up to 50 percent of those with CD4 counts < 100 cells/μL have detectable CMV DNA in plasma. CMV viraemia, even without end-organ disease, is associated with increased risk of death and opportunistic infections. However, no guidelines currently recommend antiviral therapy for CMV viraemia in this setting. International HIV guidelines emphasise early ART initiation, yet early mortality remains high irrespective of ART timing.

Valganciclovir, the oral prodrug of ganciclovir, is widely available, affordable, and effective against CMV. It has a well-characterised safety profile, though it can cause dose-related bone-marrow suppression. Observational and mechanistic studies suggest that CMV may contribute directly and indirectly to immune dysfunction, inflammation, and mortality among people with advanced HIV disease. If pre-emptive suppression of CMV replication reduces viraemia and improves outcomes, it could represent a feasible strategy to lower mortality in low-resource settings.

The NIRVANA trial will therefore assess whether valganciclovir is a safe and effective therapy for CMV viraemia in AHD. Pharmacokinetic data in this population are scarce; this study will also describe drug exposure and relationships with viral suppression and toxicity. The findings will inform the design of a larger Phase 3 trial powered to evaluate survival benefit.

Study Objectives and Hypothesis

Primary Objective:

To determine whether valganciclovir safely reduces CMV viral load compared with placebo among hospitalised adults with advanced HIV disease and CMV viraemia.

Secondary Objectives:

To assess the effect of valganciclovir on all-cause mortality and re-hospitalisation up to 12 weeks.

To characterise the pharmacokinetics of valganciclovir in this population. To evaluate tolerability and adverse-event rates. To explore immune responses, including cytokine profiles and interferon-gamma release to CMV antigen.

To describe HIV viral suppression at week 12 stratified by ART status. To examine emergence of ganciclovir resistance mutations at week 4.

Hypothesis:

Valganciclovir 900 mg once daily for 4 weeks, started at hospital admission, will significantly reduce CMV viral load compared with placebo and will be a safe therapeutic option for AHD-associated CMV viraemia.

Study Design

This is a multicentre, double-blind, parallel-group, randomised, placebo-controlled Phase 2b trial with a nested open-label pharmacokinetic sub-study. Participants meeting eligibility criteria will be randomised 1:1 to receive valganciclovir or placebo, stratified by site and baseline CMV viral load (> 1000 IU/mL). Randomisation will be implemented through a central, web-based REDCap system using computer-generated blocks to maintain allocation concealment. Study tablets for both arms are identical in appearance, packaging, and dosing schedule. Participants and all site staff involved in patient management and outcome assessment will remain blinded to allocation.

An additional non-randomised sub-study of 20 participants receiving valganciclovir will provide intensive pharmacokinetic sampling before the main randomised trial begins.

The study duration per participant is 12 weeks, including 4 weeks of study treatment and 8 weeks of post-treatment follow-up. The overall trial is expected to last approximately 24 months.

Intervention and Comparator

Experimental Arm:

Valganciclovir 900 mg once daily, taken orally for 28 days, beginning on the day of randomisation. Participants with creatinine clearance 40-60 mL/min will receive 450 mg daily.

Control Arm:

Matching placebo tablets, identical in size, colour, and packaging, administered once daily for 28 days.

All participants will continue to receive **standard of care (SOC)** for advanced HIV disease according to national or local guidelines, which may include:

Diagnosis and treatment of opportunistic infections Antiretroviral therapy (ART) initiation or re-initiation Tuberculosis preventive therapy Cotrimoxazole prophylaxis Cryptococcal antigen screening and pre-emptive antifungal therapy if positive

ART initiation will follow WHO and national recommendations, typically within 2-3 weeks of hospital admission, except for participants with cryptococcal or tuberculous meningitis, who will defer ART for 4-8 weeks.

Study Population and Setting

Study Sites:

Helen Joseph Hospital, Johannesburg, South Africa Mulago National Referral Hospital, Kampala, Uganda

Target Population:

Hospitalised adults and adolescents (≥ 15 years) with advanced HIV disease and detectable CMV viraemia.

Inclusion Criteria:

Age ≥ 15 years Confirmed HIV infection CD4 count ≤ 100 cells/µL Plasma CMV viral load > 500 IU/mL Ability to provide informed consent (or via legal surrogate if incapacitated)

Exclusion Criteria:

Clinical suspicion or diagnosis of CMV end-organ disease (including CMV retinitis) Pregnancy or breastfeeding Haematologic contraindications (absolute neutrophil count < 1.0 × 10⁹/L, haemoglobin < 8 g/dL, platelets < 100 × 10⁹/L) Estimated creatinine clearance < 40 mL/min or alanine aminotransferase > 3× upper limit of normal Current high-dose acyclovir use or concurrent myelosuppressive therapy (e.g., amphotericin B deoxycholate, linezolid) Allergy or prior adverse reaction to valganciclovir Inability to swallow tablets or expected inability to complete follow-up Moribund condition likely to result in death within 48 hours

Study Procedures and Follow-up

Screening and Consent:

All hospital admissions will be screened for HIV and CD4 count per routine care. Eligible individuals with AHD will be approached for study participation. Informed consent will be obtained in the participant's preferred language. For those lacking decision-making capacity, proxy consent from a legally authorised representative will be permitted, with re-consent sought if the participant regains capacity.

Baseline Assessments:

Demographics, clinical history, physical examination, ART status, concomitant medications, and baseline laboratory tests (haematology, renal and liver function, HIV viral load, CD4 count, CMV viral load) will be recorded in electronic case-report forms (eCRFs).

Randomisation and Treatment:

Eligible participants will be randomised via REDCap to one of the two treatment arms. Study medication will be dispensed within 24 hours of randomisation, and dosing will be supervised by nursing or study staff during hospitalisation.

Follow-up Visits:

Participants will be followed daily while in hospital, then weekly to week 4, and at weeks 8 and 12 post-randomisation. At each visit, clinical status, medication adherence, vital signs, and laboratory parameters will be reviewed. CMV viral load will be measured at baseline, days 14 and 28, and weeks 8 and 12. Blood counts, creatinine, and liver enzymes will be checked at multiple time points.

Safety Monitoring:

Adverse events of special interest (AESIs) include severe neutropenia, anaemia, thrombocytopenia, renal dysfunction, and hepatotoxicity. Participants experiencing grade ≥ 3 events will be promptly evaluated; study medication will be discontinued if no alternative cause is identified.

Pharmacokinetic (PK) Sampling:

Sparse PK samples will be collected at 2-3 hours post-dose on days 4, 7, 14, and 28 from all randomised participants. Intensive PK sampling will be performed in the sub-study cohort. Plasma samples will be analysed at the Infectious Diseases Institute laboratory in Uganda.

Immunology Sub-study:

Blood samples at baseline and selected follow-up points will be used for cytokine and interferon-gamma analyses to characterise immune response to CMV antigen.

Withdrawal and Replacement Participants discontinuing study drug will continue scheduled follow-up unless consent is withdrawn. Data collected prior to withdrawal will be retained; participants withdrawing before 4 weeks may be replaced.

Outcome Measures

Primary Outcome:

Composite of safety events (adverse events of special interest, re-hospitalisation, or death) up to 8 weeks after randomisation.

Secondary Outcomes:

Safety: same composite endpoint up to 12 weeks. Hospital length of stay post-randomisation. Serious adverse events through week 12. Mortality: survival time and all-cause mortality at 4 and 12 weeks.

Efficacy:

Median reduction in CMV viral load (log₁₀ IU/mL) from baseline to day 28 and week 12.

Proportion of participants with undetectable CMV viral load at weeks 2, 4, 8, and 12.

Tolerability: proportion of participants discontinuing study medication early. Resistance: presence of UL97 kinase or UL54 DNA polymerase gene mutations at week 4.

HIV treatment response: proportion achieving HIV RNA < 50 copies/mL at 12 weeks.

Pharmacokinetic parameters of valganciclovir. Immunologic markers of cytokine response.

Statistical Considerations

The study is powered to detect a 20 percent difference in the primary efficacy endpoint-median reduction in CMV viral load-between treatment arms with 90 percent power and a two-sided α of 0.05. Allowing for attrition, 130 randomised participants (65 per arm) will be enrolled.

Analyses will follow the intention-to-treat principle. Primary efficacy comparisons will use the geometric mean ratio of log₁₀ CMV viral load with 95 percent confidence intervals. Safety analyses will summarise adverse events by frequency and grade with absolute risk differences between arms. Missing data will be addressed using multiple imputation when appropriate. PK data will be analysed using both non-compartmental and mixed-effects modelling to explore exposure-response relationships.

Safety Monitoring and Reporting

All adverse events, serious adverse events (SAEs), and AESIs will be recorded in eCRFs. SAEs deemed related to study intervention and unexpected for the patient population will be reported promptly to the relevant institutional review boards (IRBs) and national regulatory authorities according to local requirements.

An independent Data Safety and Monitoring Committee (DSMC) will review unblinded safety and efficacy data periodically. The DSMC will include independent clinicians from Uganda and South Africa, the trial statistician, and a chairperson. Recommendations from the DSMC will guide the Trial Management Group on continuation or modification of the study.

Data Management

Data will be collected electronically using a secure REDCap platform with built-in range and consistency checks. Paper worksheets may be used temporarily if electronic capture is unavailable. The Clinical HIV Research Unit in Johannesburg will maintain the de-identified database on a secure server with restricted access. Quality-control procedures include regular data audits, query resolution, and compliance with Good Clinical Data Management Practice. Participant confidentiality will be preserved using coded identifiers; no personally identifying data will leave the site.

Ethical and Regulatory Oversight

The trial will be conducted in accordance with the principles of the Declaration of Helsinki, Good Clinical Practice (GCP), and all applicable national and institutional regulations. Ethical approval will be obtained from the University of the Witwatersrand Human Research Ethics Committee, the Uganda National Council for Science and Technology, and the London School of Hygiene and Tropical Medicine Research Ethics Committee.

Written informed consent will be obtained from all participants or their authorised representatives. Consent procedures will be conducted in participants' preferred languages, with accommodations for literacy and comprehension. All participants will be informed that participation is voluntary and that withdrawal will not affect their medical care.

Participant confidentiality will be maintained through coded data, secure storage, and controlled access. Clinical information will be released only to authorised entities such as the sponsor, IRBs, and regulatory authorities for monitoring and auditing purposes.

Study Governance

The Wits Health Consortium serves as the trial sponsor. Principal Investigators include Dr Mohammed Rassool (South Africa) and Dr Laura Nsangi (Uganda), with oversight by an international team of co-investigators from the London School of Hygiene and Tropical Medicine, the Infectious Diseases Institute (Uganda), St George's University of London, and the University of Minnesota.

A Trial Management Group (TMG) composed of investigators and the study statistician will meet regularly to monitor trial progress, review data, and approve protocol amendments and publications. An independent Trial Advisory Committee (TAC) of senior external academics will review progress approximately every six months and advise the TMG.

All investigators have completed Human Subjects Protection Training and have declared no conflicts of interest. Personnel are indemnified by their employing institutions. Funding is provided by the United Kingdom Medical Research Council.

Expected Impact

The NIRVANA trial addresses a major gap in the management of advanced HIV disease in resource-limited settings. CMV viraemia is common and strongly associated with early mortality, yet there is no evidence-based therapeutic strategy to address it. By establishing whether valganciclovir safely reduces CMV viral load and by defining its pharmacokinetics and tolerability in this population, NIRVANA will provide the essential foundation for a definitive Phase 3 trial powered to detect mortality benefit.

If successful, the findings could lead to a low-cost, implementable intervention to reduce deaths among people with advanced HIV disease worldwide.

ELIGIBILITY:
Inclusion Criteria:

Confirmed HIV infection CD4 count ≤100 cells/mm³ Expected to survive at least 48 hours CMV viral load >500 international units (IU) / mL in blood. Provision of informed consent

Exclusion Criteria:

Confirmed or high level of clinical suspicion for CMV end organ disease as determined by the treating team CMV retinitis confirmed by retinal phography Pregnancy or breastfeeding Contraindication to valganciclovir (absolute neutrophil count < 1.0 X109/L, haemoglobin < 8 g/dL, platelets < 100 X109/L) Allergy or prior adverse reaction to valganciclovir Expected to be unable to complete follow up Moribund - treating team considers patient is likely to die within next 48 hours Estimated creatinine clearance < 40 mL/min ALT > 3X ULN Receipt of high dose acyclovir as standard of care Unable to swallow whole tablets Concurrent administration of highly myelosuppressive drug, e.g. amphotericin B deoxycolate and linezolid

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events of special interest plus re-hospitalisation or death up to week 8 | 8 weeks post randomisation
  Adverse Events of Special Interest• Absolute neutrophil count < 0.4 X109/L
  * Haemoglobin < 7 g/dL
  * Platelets < 50 X109/L
  * Creatinine increases to > 1.5X participant's baseline
  * ALT > 5X ULN

IPD SHARING:
Plan to Share IPD: Yes
All
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: August 2027 to July 2030
Access Criteria: Reputable researchers